CLINICAL TRIAL: NCT06281275
Title: A Study on the Association Between Frailty and Acute Postoperative Pain in Elderly Patients Undergoing Thoracoscopic Surgery and an Investigation of the Mechanisms Involved
Brief Title: A Study of the Association Between Frailty and Acute Postoperative Pain in Elderly Thoracoscopic Surgery Patients
Status: Recruiting | Type: Observational
Sponsor: Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Xianwei Zhang，MD, Clinical Professor, Huazhong University of Science and Technology
Other Study IDs: TJ-IRB202402008
Record Dates: First submitted 2024-02-20; First posted 2024-02-28 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-06

CONDITIONS: Frailty; Acute Postoperative Pain
Keywords: Frailty; Acute Postoperative Pain; Gastrointestinal Microbiome; Thoracoscopy
MeSH Terms: conditions — Frailty; Pain, Postoperative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 1. Purpose Before the start of this study, we obtained consent from the subjects to collect fecal samples and blood samples and to use these samples for the analysis of intestinal flora and biochemical indices.
  2. Sample type and purpose Stool samples: To analyze the composition of the intestinal flora. Blood samples: for the detection of inflammatory factors and oxidative stress.
  3. Harmonized storage and destruction Preservation: All samples will be preserved after collection to ensure security and data confidentiality.
  Destruction Policy: All samples will be securely destroyed at the end of the study to ensure personal data security and compliance with ethical requirements.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To gain a clearer understanding of the association between frailty and postoperative acute pain in elderly thoracoscopic surgery patients and its underlying mechanisms, to provide new solution ideas to reduce the level of postoperative acute pain and improve the debilitating state of elderly thoracoscopic surgery patients, and consequently improve their quality of life and mental status.

DETAILED DESCRIPTION:
Frailty, as a geriatric syndrome, is recognized as being characterized by a decline in the reserve capacity of the body's physiological systems1 and, in severe cases, by regulatory disorders, which result in a decrease in the individual's resistance and resilience to a variety of contingency sources, including organismal, physiological, and psychological stressors as well as an increase in organismal susceptibility to damage. The globe is accelerating its entry into an aging society, and, according to the World Health Organization's report on aging and health reports, the proportion of the world's population over the age of 60 will increase from 12% to 22% between 2015 and 2050. As the population ages, the prevalence of frailty in healthy populations increases exponentially with age. The prevalence in healthy populations ranges from 6.5% in healthy people between the ages of 60-69 years to as high as 65% or even higher in healthy people over the age of 85 years. The prevalence of frailty in healthy populations has been shown to increase with age.

Frailty is now an emerging global health burden, with a meta-analysis of studies from 62 countries noting a 24% prevalence of frailty and a 49% prevalence of pre-frailty in people over the age of 50. Frailty typically prolongs hospital stays and increases hospitalization costs for older patients, increases the prevalence of depression and the risk of cardiovascular disease, increases intraoperative blood loss in patients, and even leads to an increased risk of new-onset disability and death in individuals. Frailty has been shown to increase the risk of new-onset disability, death in individuals, and intraoperative blood loss in patients. Frailty can even lead to an increased risk of new-onset disability and death in individuals.

Currently, the proportion of elderly patients undergoing surgery is also increasing. With the development of minimally invasive surgery, more and more thoracic surgical diseases are treated with thoracoscopic surgery, which is characterized by smaller incisions, less trauma, better results, and the promotion of rapid recovery, compared with open thoracic surgery. Despite the rapid and minimally invasive development of thoracic surgery, postoperative pain after lung surgery is severe, and patients in the first few hours after surgery may still experience severe pain. Postoperative pain can lead to adverse consequences such as decreased quality of life and impact on physical and mental health. Some studies have shown that older adults with early-onset debility have a high prevalence of chronic pain, and risk factors for the development of debility include the prolonged presence of pain. Thus, there may be an unproven bidirectional relationship between debility and pain.

Currently, the mechanisms of the development of frailty are unknown, and Frailty is associated with gut microbiota and biomarkers. Therefore, a clear understanding of the association between frailty and acute postoperative pain in elderly thoracoscopic surgery patients and its underlying mechanisms is essential to reduce the level of acute postoperative pain and improve the frailty status of elderly thoracoscopic surgery patients, but also important to improve their quality of life and mental status.

ELIGIBILITY:
Inclusion Criteria:

1. patients undergoing thoracic surgery under general anesthesia with 48 h of postoperative patient-controlled analgesia;
2. age ≥60 years;
3. ASA class I-III;
4. signed informed consent;
5. patients undergoing thoracoscopic surgery.

Exclusion Criteria:

1. Patients who themselves refuse to participate in the study;
2. Drug dependence;
3. Patients who cannot cooperate with communication and have verbal communication difficulties;
4. Patients who cannot assess frailty preoperatively and pain postoperatively;
5. Failure to provide a compliant fecal sample at the agreed time;
6. antibiotic treatment within the last month;
7. intestinal dysfunction (e.g., irritable bowel syndrome, inflammatory bowel disease, chronic diarrhea, and other types of intestinal disorders);
8. comorbidities of certain metabolic disorders (e.g., thyroid dysfunction, diabetes mellitus, and so on) that may affect the structure of the microbial community;

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: It is proposed to observe cases with age greater than or equal to 60 years undergoing thoracoscopic surgery at Tongji Hospital from February 2024 to October 2024 who meet the inclusion and exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 78 (Estimated)
Dates: Start 2024-03-12 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-10-30 (Estimated)

PRIMARY OUTCOMES:
All patients' Numerical Rating Scale （NRS） scores for most significant pain at rest in the 48h postoperative period | 202402-2024-10
  Patients' pain levels were assessed using the Numerical Rating Scale （NRS） scale. This method is composed of a total of 11 numbers from 0 to 10, the patient with 0 to 10 of these 11 numbers to describe the intensity of pain, the greater the number of pain is increasingly serious. 0 no pain, 1 to 3 mild pain (pain does not affect sleep), 4 to 6 moderate pain, 7 to 6 pain is increasingly serious. The patient describes the intensity of pain using the 11 numbers from 0 to 10, the greater the number, the more severe the pain becomes. 0 no pain, 1-3 mild pain (pain that does not interfere with sleep), 4-6 moderate pain, 7-9 severe pain (inability to sleep or waking up from sleep with pain), and 10 severe pain.
Numerical Rating Scale （NRS） scores for the most pronounced pain in the patient's coughing state in the 48h postoperative period | 202402-2024-10
  All patients' pain levels were assessed using the NRS scale. This method is composed of a total of 11 numbers from 0 to 10, the patient with 0 to 10 of these 11 numbers to describe the intensity of pain, the greater the number of pain is increasingly serious. 0 no pain, 1 to 3 mild pain (pain does not affect sleep), 4 to 6 moderate pain, 7 to 6 pain is increasingly serious. The patient describes the intensity of pain using the 11 numbers from 0 to 10, the greater the number, the more severe the pain becomes. 0 no pain, 1-3 mild pain (pain that does not interfere with sleep), 4-6 moderate pain, 7-9 severe pain (inability to sleep or waking up from sleep with pain), and 10 severe pain.

SECONDARY OUTCOMES:
PCA pump consumption | 202402-2024-10
  All patients' pain levels were assessed using the Numerical Rating Scale （NRS）, which is composed of a total of 11 numbers from 0 to 10, the patient with 0 to 10 of these 11 numbers to describe the intensity of pain, the greater the number of pain is increasingly serious. 0 no pain, 1 to 3 mild pain (pain does not affect sleep), 4 to 6 moderate pain, 7 to 6 pain is increasingly serious. The patient describes the intensity of pain using the 11 numbers from 0 to 10, the greater the number, the more severe the pain becomes. 0 no pain, 1-3 mild pain (pain that does not interfere with sleep), 4-6 moderate pain, 7-9 severe pain (inability to sleep or waking up from sleep with pain), and 10 severe pain.
Number of PCA pump presses | 202402-2024-10
  Check the analgesic pump and record the number of active analgesic pump compressions

CONTACTS AND LOCATIONS:
Overall Officials: Xianwei Zhang, Doctor, Principal Investigator — Huazhong University of Science and Technology
Locations (1):
- Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Tanaka S, Kamiya K, Matsue Y, Yonezawa R, Saito H, Hamazaki N, Matsuzawa R, Nozaki K, Yamashita M, Wakaume K, Endo Y, Maekawa E, Yamaoka-Tojo M, Shiono T, Inomata T, Ako J. Efficacy and Safety of Acute Phase Intensive Electrical Muscle Stimulation in Frail Older Patients with Acute Heart Failure: Results from the ACTIVE-EMS Trial. J Cardiovasc Dev Dis. 2022 Mar 27;9(4):99. doi: 10.3390/jcdd9040099. PMID 35448075
- [Background] Miyano T, Kaneko R, Kimura T, Maruoka M, Kishimura A, Kato K, Furuta M, Yamashita Y. Dietary Problems Are Associated with Frailty Status in Older People with Fewer Teeth in Japan. Int J Environ Res Public Health. 2022 Dec 5;19(23):16260. doi: 10.3390/ijerph192316260. PMID 36498332
- [Background] Morley JE, Vellas B, van Kan GA, Anker SD, Bauer JM, Bernabei R, Cesari M, Chumlea WC, Doehner W, Evans J, Fried LP, Guralnik JM, Katz PR, Malmstrom TK, McCarter RJ, Gutierrez Robledo LM, Rockwood K, von Haehling S, Vandewoude MF, Walston J. Frailty consensus: a call to action. J Am Med Dir Assoc. 2013 Jun;14(6):392-7. doi: 10.1016/j.jamda.2013.03.022. PMID 23764209
- [Background] Gale CR, Cooper C, Sayer AA. Prevalence of frailty and disability: findings from the English Longitudinal Study of Ageing. Age Ageing. 2015 Jan;44(1):162-5. doi: 10.1093/ageing/afu148. Epub 2014 Oct 12. PMID 25313241
- [Background] O'Caoimh R, Sezgin D, O'Donovan MR, Molloy DW, Clegg A, Rockwood K, Liew A. Prevalence of frailty in 62 countries across the world: a systematic review and meta-analysis of population-level studies. Age Ageing. 2021 Jan 8;50(1):96-104. doi: 10.1093/ageing/afaa219. PMID 33068107
- [Background] Lakra A, Tram MK, Bernasek TL, Lyons ST, O'Connor CM. Frailty is Associated With Increased Complication, Readmission, and Hospitalization Costs Following Primary Total Knee Arthroplasty. J Arthroplasty. 2023 Jul;38(7 Suppl 2):S182-S186.e2. doi: 10.1016/j.arth.2023.02.036. Epub 2023 Feb 28. PMID 36858131
- [Background] Gu C, Lu A, Lei C, Wu Q, Zhang X, Wei M, Wang Z. Frailty index is useful for predicting postoperative morbidity in older patients undergoing gastrointestinal surgery: a prospective cohort study. BMC Surg. 2022 Feb 16;22(1):57. doi: 10.1186/s12893-022-01471-9. PMID 35172806
- [Background] Fluitman KS, Davids M, Olofsson LE, Wijdeveld M, Tremaroli V, Keijser BJF, Visser M, Backhed F, Nieuwdorp M, IJzerman RG. Gut microbial characteristics in poor appetite and undernutrition: a cohort of older adults and microbiota transfer in germ-free mice. J Cachexia Sarcopenia Muscle. 2022 Aug;13(4):2188-2201. doi: 10.1002/jcsm.13002. Epub 2022 Jun 14. PMID 35698917